CLINICAL TRIAL: NCT00726700
Title: Randomized Phase II Study About the Application of Pegfilgrastim (Neulasta) at Day 2 or Day 4 Within the Treatment in Patients With Aggressive Non-Hodgkin's Lymphoma Aged 61 to 80 Years With 6 or 8 Cycles of Chemotherapy With CHOP (Cyclophosphamide, Doxorubicin, Vincristine and Prednisone) at 14-day Intervals (CHOP-14), Both With or Without the Monoclonal Anti-CD20 Antibody Rituximab
Brief Title: Pegfilgrastim and Combination Chemotherapy With or Without Rituximab in Treating Older Patients With Aggressive B-Cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: DSHNHL-2003-2; CDR0000454473 (Registry Identifier: PDQ (Physician Data Query)); EU-20534
Record Dates: First submitted 2008-07-31; First posted 2008-08-01 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Lymphoma
Keywords: stage III grade 3 follicular lymphoma; stage I adult lymphoblastic lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; anaplastic large cell lymphoma; stage III adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; stage III mantle cell lymphoma; stage I mantle cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage I adult Burkitt lymphoma; contiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult Burkitt lymphoma; stage III marginal zone lymphoma; stage IV marginal zone lymphoma; stage I marginal zone lymphoma; contiguous stage II marginal zone lymphoma; noncontiguous stage II marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — pegfilgrastim; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

ARMS (2):
- Arm I (without rituximab) (Active Comparator): Patients receive pegfilgrastim subcutaneously (SC) on day 2 or 4 and CHOP comprising cyclophosphamide IV, doxorubicin IV, vincristine IV on day 1, and oral prednisone on days 1-5. Treatment repeats every 2 weeks for up to 6-8 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: pegfilgrastim; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate
- Arm II (with rituximab) (Experimental): Patients receive pegfilgrastim and CHOP for up to 6-8 courses as in arm I. They also receive rituximab (administered 2 hours before beginning CHOP) on day 1. Treatment with rituximab repeats every 2 weeks for up to 8 courses.
  Interventions: Biological: pegfilgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate

INTERVENTIONS:
Biological: pegfilgrastim — Given subcutaneously
Biological: rituximab — Given IV
  Arms: Arm II (with rituximab)
Drug: cyclophosphamide — Given IV
Drug: doxorubicin hydrochloride — Given IV
Drug: prednisone — Given orally
Drug: vincristine sulfate — Given IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, and vincristine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Colony-stimulating factors, such as pegfilgrastim, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. It is not yet known whether combination chemotherapy and pegfilgrastim is more effective when given with or without rituximab in treating non-Hodgkin lymphoma.

PURPOSE: This phase II trial is studying the side effects of giving pegfilgrastim and combination chemotherapy together with or without rituximab and to see how well it works in treating older patients with aggressive B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the side effects of pegfilgrastim and cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone (CHOP) with or without rituximab in older patients with aggressive B-cell non-Hodgkin lymphoma.
* Determine adherence to therapy regimens in these patients.
* Determine antitumor effectivity of immunochemotherapy.

OUTLINE: This is a multicenter study.

All patients receive prephase treatment comprising vincristine on day -6 and prednisone on days -6 to 0. Patients are then randomized to 1 of 2 treatment arms.

* Arm I (without rituximab): Patients receive pegfilgrastim subcutaneously (SC) on day 2 or 4 and CHOP comprising cyclophosphamide IV, doxorubicin hydrochloride IV, and vincristine IV on day 1, and oral prednisone on days 1-5. Treatment repeats every 2 weeks for up to 6-8 courses in the absence of disease progression or unacceptable toxicity.
* Arm II (with rituximab): Patients receive pegfilgrastim and CHOP for up to 6-8 courses as in arm I. They also receive rituximab (administered 2 hours before beginning CHOP) on day 1. Treatment with rituximab repeats every 2 weeks for up to 8 courses.

Patients with bulky disease or extranodal disease also undergo radiotherapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of CD20-positive B-cell non-Hodgkin lymphoma (NHL)

  * Confirmed by an excisional biopsy of a lymph node or by a sufficiently extensive biopsy of an extranodal involvement (if there is no lymph node involvement)
  * Results of the immunohistological analysis of expression of the CD20 antigen by lymphoma cells must be obtained
* Aggressive disease, including any of the following B-cell NHL

  * Stage III follicular lymphoma
  * Stage III follicular lymphoma and diffuse B-cell lymphoma
  * Lymphoblastic precursor B-cell lymphoma
  * Diffuse large B-cell lymphoma, including any of the following subtypes:

    * Centroblastic
    * Immunoblastic
    * Plasmablastic
    * Anaplastic large cell
    * T-cell rich B-cell lymphoma
    * Primary effusion lymphoma
    * Intravasal B-cell lymphoma
    * Primary mediastinal B-cell lymphoma
  * Mantle zone lymphoma
  * Burkitt or Burkitt-like lymphoma
  * Aggressive marginal zone lymphoma (monocytoid)
* All risk group allowed

  * Age adjusted IPI 0-3
* Previously untreated disease

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* No other serious concurrent diseases

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 61 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2004-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
comparison of pegfilgrastim day 4 versus day 2 for the prevention of chemotherapy-induced leukocytopenia | through chemotherapy administration (up to 112 days respectively)
  median of two measurements of hemoglobin, leukocyte and platelet counts per chemotherapy cycle per Patient in correlation with median pegfilgrastim serum levels at day 1 of the next chemotherapy cycle
comparison of pegfilgrastim day 4 versus day 2 for the prevention of chemotherapy-induced leukocytopenia | through chemotherapy administration (up to 112 days respectively)
  rates and grades of leukocytopenias and infections according to NCI-CTC criteria (version 2)

SECONDARY OUTCOMES:
Adherence to therapy regimens | through chemotherapy administration (up to 112 days respectively)
  the median overall treatment duration
Antitumor effectivity | median time of observation up to 3 years
  progression-free survival
Disease-free survival | median time of observation up to 3 years
  period of disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hartmann, MD, Study Chair — Universitaetsklinikum des Saarlandes

REFERENCES:
- [Background] Zwick C, Hartmann F, Zeynalova S, Poschel V, Nickenig C, Reiser M, Lengfelder E, Peter N, Schlimok G, Schubert J, Schmitz N, Loeffler M, Pfreundschuh M; German High-Grade Non-Hodgkin Lymphoma Study Group. Randomized comparison of pegfilgrastim day 4 versus day 2 for the prevention of chemotherapy-induced leukocytopenia. Ann Oncol. 2011 Aug;22(8):1872-7. doi: 10.1093/annonc/mdq674. Epub 2011 Feb 3. PMID 21292644
- [Derived] Muller C, Murawski N, Wiesen MH, Held G, Poeschel V, Zeynalova S, Wenger M, Nickenig C, Peter N, Lengfelder E, Metzner B, Rixecker T, Zwick C, Pfreundschuh M, Reiser M. The role of sex and weight on rituximab clearance and serum elimination half-life in elderly patients with DLBCL. Blood. 2012 Apr 5;119(14):3276-84. doi: 10.1182/blood-2011-09-380949. Epub 2012 Feb 15. PMID 22337718
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21292644/